CLINICAL TRIAL: NCT05452343
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Subjects With Chronic Pruritus of Unknown Origin
Brief Title: A Study of CM310 in Subjects With Chronic Pruritus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310_IIS_CP02
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pruritus of Unknown Origin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 (Experimental): 600 mg (first dosing) + 300 mg (subsequent dosing), once every two weeks
  Interventions: Biological: CM310
- Placebo (Placebo Comparator): once every two weeks
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — 600 mg (first doing) + 300 mg (subsequent dosing), once every two weeks

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled Phase II study to evaluate the efficacy and safety of CM310 in subjects with chronic pruritus of unknown origin.

DETAILED DESCRIPTION:
The study consists of a Screening Period (up to 4 weeks), Treatment Period (16 weeks) and Safety Follow-up Period (8 weeks).

50 subjects who meet eligibility criteria will be randomized 1:1 to receive either CM310 300 mg or matched placebo subcutaneously every two weeks (Q2W) for a total of 8 times. All subjects will receive mometasone furoate nasal spray (MFNS) on a daily basis as a background treatment throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* With chronic pruritus of unknown origin.
* With the worst pruritus numerical rating scale (WI-NRS) ≥7.
* Contraception.

Exclusion Criteria:

* Heavy drinking in the 3 months prior to screening.
* With severe hepatic and renal impairment.
* Previous history of autosensitivity dermatitis.
* Allergic to CM310/placebo.
* Vaccination with live attenuated vaccine within 12 weeks before randomization or during the planned study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change of weekly average in the worst itching numerical rating scale (WI-NRS) | at week 16
  Change from baseline in the worst itching numerical rating scale at week 16

SECONDARY OUTCOMES:
Safety parameters | Baseline up to Week 24
  Incidence of treatment-emergent adverse events (TEAEs).